CLINICAL TRIAL: NCT00208221
Title: Comparison of a Higher Dose of Ramipril to the Addition of Telmisartan 80 mg+Ramipril 10 mg in Patients With Hypertension and Diabetes
Brief Title: Higher Dose of Ramipril Versus Addition of Telmisartan-Ramipril in Hypertension and Diabetes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Not enough recruitment
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RD 0507/17259
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-11-08 (Estimated); Status verified 2007-11

CONDITIONS: Hypertension; Type 2 Diabetes; Albuminuria
Keywords: Hypertension; Diabetes; Microalbuminuria; Blood pressure
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Albuminuria; Diabetes Mellitus | interventions — Ramipril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ramipril
Drug: ramipril-telmisartan

SUMMARY:
The purpose of this study is to determine if a dose of ramipril combined with a normal dose of telmisartan 80 mg will be more effective than ramipril 20 mg in reducing microalbuminuria in hypertensive patients with diabetes.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of ramipril 10 mg and telmisartan 80 mg versus ramipril 20 mg in patients with diabetes type II, hypertension and microalbuminuria (Urinary-albuminuria creatinine ratio of 2.0 to 25 mg/mmol) on

1. Microalbuminuria
2. Blood pressure (systolic, diastolic and ABPM), Renin-angiotensin system, Catecholamines, Oxydative stress
3. Comparison at 4, 8 and 12 weeks with addition of hydrochlorothiazide 12.5 mg if BP over 130/80 mmHg

ELIGIBILITY:
Inclusion Criteria:

* Male or female over the age of 18 years
* Diastolic blood pressure (DBP) greater tha 80 mmHg and less than 104 mmHg
* Type II diabetes on diet or oral hypoglycemic agents with a hemoglobin A1C (HbA1C) less than 0.080
* UA ratio albumin:creatinine 2.0 to 25 mg/mmol

Exclusion Criteria:

* DBP > 104 mmhg
* Woman not surgically sterile or menopausal.
* Premenopausal women whoo are not surgically sterile or who are not practicing acceptable means of birth control and do not agree to submit to periodic pregnancy tests.
* Known or secondary forms of hypertension.
* Intolerance to angiotensin (AT) 1 receptor blockers or angiotensin-converting enzyme (ACE) inhibitors.
* Hepatic or renal dysfunction. Creatinine > 150 umol or enzymes greater than 2 times upper limit of normal.
* Hemodynamically significant renal artery stenosis, renal artery stenosis on a solitary kidney, post-renal transplant or with only one kidney.
* Uncorrected volume depletion.
* Biliary obstructive disorders.
* NYHA functional class congestive heart failure (CHF) III-IV.
* Coronary heart disease needing pharmacological therapy.
* Stroke within the preceding six months.
* Percutaneous transluminal coronary angioplasty (PTCA) within the preceding three months.
* History of angioedema.
* Sustained ventricular tachycardia, atrial fibrillation, or other clinically relevant cardiac arrhythmias as determined by the clinical investigator.
* Second or third degree AV block, left bundle branch block or any clinically relevant conduction abnormality as determined by the clinical investigator.
* Hypertrophic obstructive cardiomyopathy, aortic stenosis, hemodynamically relevant stenosis of aortic or mitral valve.
* Administration of digoxin.
* Patients with a fasting glucose greater than 7.0
* History of drug or alcohol dependency.
* Use of antihypertensive agents such as diuretics, ACE inhibitors, angiotensin II antagonists, alpha-blockers, beta-blockers, calcium channel antagonists, direct vasodilators that cannot be stopped for the trial.
* Administration of other non-antihypertensive medications known to affect blood pressure (e.g. oral corticosteroids, monoamine oxidase [MAO] inhibitors, nitrates) at any time during the trial.
* Chronic use of salt substitutes containing potassium chloride; potassium supplements; extreme dietary restrictions.
* Uncorrected sodium depletion as defined by a serum sodium level less than 135 mEq/L.
* Clinically significant hyperkalemia as defined by serum potassium level greater than 5.2 mEq/L. Clinically significant hypokalemia as defined by serum potassium level less than 3.0 mEq/L.
* Patients receiving any investigational therapy within one month of signing the informed consent form.
* Known hypersensitivity to any component of telmisartan, ramipril or hydrochlorothiazide.
* Any other clinical condition which, in the opinion of the principal investigator, would not allow safe completion of the protocol and safe administration of trial medication.
* Blood donation in the preceding 1 month.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-08; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Microalbuminuria

SECONDARY OUTCOMES:
Plasma renin
plasma angiotensin
plasma aldosterone
plasma catecholamines
oxydative stress
diastolic blood pressure
systolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Larochelle, MD PhD FRCPC, Principal Investigator — Institut de Recherches Cliniques de Montreal
Locations (1):
- Institut de Recherches Cliniques de Montreal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Natale P, Palmer SC, Navaneethan SD, Craig JC, Strippoli GF. Angiotensin-converting-enzyme inhibitors and angiotensin receptor blockers for preventing the progression of diabetic kidney disease. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD006257. doi: 10.1002/14651858.CD006257.pub2. PMID 38682786